CLINICAL TRIAL: NCT02017873
Title: "Evaluation of the Effectiveness and Longevity Post Whitening Carbamide Peroxide 10% in Smokers and Nonsmokers. Double-blind Multicenter Clinical Trial. "
Brief Title: Longevity and Effectiveness of Bleaching in Healthy and Smokers Patients
Acronym: BLESMOK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Eduardo Maximiliano Fernández Godoy, University of Chile
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nº 2013/41 FOUCH
Record Dates: First submitted 2013-12-05; First posted 2013-12-23 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Dentin Sensitivity
Keywords: bleaching; smokers; effectiveness; pain
MeSH Terms: conditions — Dentin Sensitivity; Pain | interventions — Carbamide Peroxide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- healthy patients bleaching (Active Comparator): Healthy patients Peroxide Carbamide 10% - Dental bleaching treatment
  Interventions: Drug: Peroxide Carbamide 10% - Dental bleaching treatment
- Smokers bleaching (Experimental): smokers patients Peroxide Carbamide 10% - Dental bleaching treatment
  Interventions: Drug: Peroxide Carbamide 10% - Dental bleaching treatment

INTERVENTIONS:
Drug: Peroxide Carbamide 10% - Dental bleaching treatment — During 3 hours in 3 weeks of bleaching in both groups in healthy patients and smokers patients
  Other Names: FGM Peroxide Carbamide ( Joinville , Brazil )

SUMMARY:
The main objective of this study is to evaluate the effectiveness and longevity of color and Tooth sensitivity of patients undergoing home whitening peroxide 10% carbamide ( Whiteness Perfect , FGM , Joinville , Santa Catarina , Brazil) , and the relationship with the cigarette use for tooth whitening. They will be selected 120 patients with incisors darker than A2, higher plants will be divided into 2 groups per center (n = 30 ) , GE - Group Experimental ( smoking) and GC - Group Control ( non-smoking) . For the two groups will be used Carbamide peroxide 10% for 3 hours daily for a period of 3 weeks. Color will evaluated through the Vita Classical scale and Vita Easyshade Spectrophotometer in the periods: Home , for tooth whitening (1st , 2nd and 3rd week) and post- whitening ( 1 week and 1 month , 2 and 3 months). Patients recorded the perceived sensitivity through Numerical Analogue Scale (NRS ) with values from 0 to 4, where 0 = no sensation, 1 = mild, 2 = moderate, 3 = severe and 4 = significant , also in the Visual Analogue Scale (VAS ), with values from 0 to 10 where 0 = 10 = severe tenderness and sensitivity. for color analysis will be made two-way ANOVA (group vs. treatment time ), being Over time the repeated measure ( α = 0.05). Test will be held on Tukey to contrast the average ( α = 0.05). The sensitivity will be evaluated by the Fisher exact test . It is expected that there is no difference on the effectiveness of home whitening and tooth sensitivity between smokers and nonsmokers.

DETAILED DESCRIPTION:
This study will be conducted under the CONSORT recommendations and respecting the principles of Helsinsky convention and corresponds to a multicenter study in conjunction with the University of Ponta Grossa Brazil (Deputy resolution protocol and ethics committee (Appendix A and B ) . Will be invited to participate in the study to patients who come to the clinic through FOUCH public posters. Subsequently 120 volunteers will be selected on the criteria that qualify inclusion and exclusion from the study will be reported all volunteers were examined not qualify under the criteria for inclusion as part of the initial n , according to CONSORT recommendations .

After signing the informed ( TCLE ) consent (Appendix 3 ) shall be made prophylaxis teeth of the upper and lower teeth , for the removal of extrinsic stains jet sodium bicarbonate ( Profi class , Ribeirao Preto , Sao Paulo , Brazil) , two weeks before the beginning of tooth whitening.

Inclusion and exclusion criteria:

Patients included in this study must be over 18, in good general health and buccal, have teeth free of carious lesions and periodontal disease, which agree with the informed consent document . And the color of the anterior teeth higher is classified as A2 or greater value , according to the scale VITA Classical (Vita Zahnfabrik, Bad Sackingen, Germany) and the spectrophotometer Easyshade Vita (Vita Zahnfabrik, Bad Sackingen, Germany). Evaluation of color through the VITA scale Classical will be made independently by two calibrated investigators and blind.

Be excluded from the study patients: they have already made treatment tooth whitening, or dental prosthesis having options at the upper front teeth , who are pregnant or lactating , presenting gingival recession, sensitivity dental, endodontic treatment in anterior maxillary teeth, which have a coloring severe internal, if they have non-carious cervical lesions, are taking medications , using fixed orthodontic appliances, submit bruxism habits, which have visible teeth cranks and those who are not available to attend the controls.

Study Design Patients will be divided into two groups (n = 60 ), GC (control group) and GE (group experimental ). At the initial consultation volunteers will be asked about smoking habits daily. Patients who do not smoke will be part of the GC, and heavy smokers (more than 10 day ) will be part of GE.A cigarettes all smokers are complementary be given a booklet of tips for quitting smoking and damage, and sites where to find more information. (Annex C ) The teeth whitening technique selected for this study, is the technique of home bleaching, validated for both groups. Treatment and follow-up will no cost to the patient . For the development of individual buckets, this will be through impression of the upper and lower arch of each patient Jeltrate Plus alginate ( Dentply, Petrópolis, Rio de Janeiro, Brazil), the molds will be cast in plaster and immediately after printing. After obtaining this plaster model is cut and taken to the vacuum laminator ( Protécni, Araraquara, Sao Paulo, Brazil) for making buckets individual vinyl acetate 1 mm thick (Plate Pail Whiteness -FGM, Joinville, Santa Catarina, Brazil). Cuvettes acetate be cut an inch margin on gingival . For both groups of PC gel will be used 10% ( Whiteness Perfect, FGM, Joinville, Santa Catarina, Brazil ), for a period of 3 hours a day for three weeks ) . After the test cuvette acetate individual, the method of application of the product will be carefully explained to each patient in the study as follows : Dispense a drop in the region of the product corresponding to the buccal surface of each tooth in the tray. The amount of gel should be sufficient to remain in contact with the buccal tooth surface without covering the gingival third, preventing injuries from it. After this period, patients will be instructed to withdraw the tray with the whitening gel and perform vigorous mouth rinsed with water to complete removal of the product.

Evaluation of Color Subjective method Color will be assessed by the scale VITA Classical (Vita Zahnfabrik, Bad Sackingen, Germany ), consisting of 16 color guides, organized by value, higher value (B1 ) to low value ( C4 ). Although this scale is not linear, it is organized according to a ranking range valor. Represent and the purpose of analysis.

Two blind reviewers record the color of the right maxillary central incisor patients through the scale VITA Classical (Vita Zahnfabrik, Bad Sackingen, Germany). At the following times : initial, 1st week, 2nd week, 3rd week (active phase bleaching) and post- bleaching periods : 1 week, 1 month, 2 and 3 months. Evaluators always record the color independently in the same room with the same lighting. If there is a discrepancy in the color registration, a new evaluation will be conducted together until a consenso. The area chosen for color measurement is the middle third of the labial surface of the central incisor, according to the ADA specifications . The color change will be evaluated by means of varying scale Vita units ( ΔUEV ) organized by value.

Objective method The color will also be measured with the spectrophotometer Easyshade ( Vita Zahnfabrik, Bad Sackingen, Germany ) according to the CIELab system of Vita. Calibration of equipment will always be made before each measurement, and three measurements for each tooth will be made. The evaluation will be conducted at the same times that the method subjective. For standardize the measuring of color, a mold of the teeth of the upper arch with heavy condensation silicone (Coltoflax profile and cub, Vigodent, Rio de Janeiro will be held, Brazil ) for making a silicone matrix. The matrix was used to standardize the region of the tooth in which the color is measured with the spectrophotometer. The matrix will be drilled in the vestibular region, in the middle third, in the upper teeth, using a scalpel circular 6 mm in diameter, Biopsy punch ( Miltex, York, PA USA), similar diameter to the tip of the spectrophotometer Vita Easyshade. Color recurrence begins the day the patient is bleached, the spectrophotometer used has a sufficient sensitivity to determine minimal color changes, is based on the construction algorithm for the detection of the dimensions h and b color . (Jadad et al. , 2011)

Evaluation of the Dental Sensitivity In the initial clinical examination of patients , baseline sensitivity is measured by the vertical , horizontal drum , air jet application and probing of all teeth, so it can be compared with the sensitivity during the whitening dental.Durante whitening, patients record the presence or absence of tooth sensitivity, in a newspaper of tooth sensitivity using analog numerical scale (ENR ), with values from 0 to 4, where: 0 = no tenderness, 1 = Slight, 2 = moderate 3 = considerably and 4 = severe. And on the visual analogue scale (VAS ) with values from 0 to 10 where 0 = no sensitivity and 10 = severe. Patients mark a vertical line across the horizontal line of the scale corresponding to the intensity of tooth sensitivity. After measurement in millimeters are made with the aid of a millimeter ruler. Annex 5 and 6 values will be organized into two categories: percentage of patients with tooth sensitivity at some time during treatment ( absolute risk sensitivity ) and intensity of tooth sensitivity.

Patients with severe sensitivity will be immediately assisted by investigators to reverse the painful picture using desensitizing and / or analgesics and anti-inflammatories for pain relief, the patient will be removed from study. If sensitivity is used desensitizing FMG KF 2% ( nitrate Potassium and Sodium Fluoride 2%, Joinville, Brazil) , the literature does not present any report about RAM, if for any reason there is any Medical Adverse Event the research team will be responsible for any additional medical or dental treatment required and its follow-up, in the wake of whitening procedure ( restorations, endodontics, etc. )

Statistical Analysis The color data obtained by the objective and subjective analysis will be evaluated by analysis of variance of two factors (ANOVA ) for repeated measures ( time vs. treatment groups ) ( α = 0.05). Tukey's test performed to test the means ( α = 0.05). The absolute risk of sensitivity will be evaluated by the Fisher exact test .

Sampling calculation was obtained by the G -Power 3.1 program considering a Beta error 0.8, and an alpha error 0.05, meaning a sample calculation of 25 patients per group per center, considering the drop-out reported in other published work ( 5%) was decided to increase to 30 the n sample size for each group per center. Coincident with the Odds Ratio of all clinical work whitening the past 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study must be over 18 years with good general and oral health
* Free teeth having carious lesions and periodontal disease agree with the informed consent document
* The color of the upper anterior teeth is classified as A2 or greater value, according to the scale VITA Classical (Vita Zahnfabrik, Bad Sackingen, Germany) and the spectrophotometer Easyshade Vita (Vita Zahnfabrik, Bad Sackingen, Germany).

Exclusion Criteria:

* Have already made treatment tooth whitening
* Dental prosthesis having options at the upper front teeth
* Who are pregnant or lactating
* Presenting gingival recession
* Tooth sensitivity
* Endodontic treatment in anterior maxillary teeth
* Which have a severe internal coloring
* Cervical lesions carious
* Taking medications (AINES)
* Fixed orthodontic appliances
* Submit bruxism habits
* Having visible cracks in teeth
* Those who are not available to attend the controls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Color | 1, 2, 3, 4, 8 weeks and 3, 6, 9 and 12 month
  Objective ( Vita Easy shade ), Subjective measurement

SECONDARY OUTCOMES:
Sensitivity | 1, 2, 3, 4, 8 weeks 3, 6, 9,12 month
  VAS Scale 0-4 Pain Scale

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fernandez, Prof., Principal Investigator — University of Chile
Locations (2):
- Juliana Larocca de Geus, Ponta Grossa, Brazil
- Faculty of Dentistry - University of Chile, Santiago, Metropólitana, Chile

REFERENCES:
- [Background] de Geus JL, Bersezio C, Urrutia J, Yamada T, Fernandez E, Loguercio AD, Reis A, Kossatz S. Effectiveness of and tooth sensitivity with at-home bleaching in smokers: a multicenter clinical trial. J Am Dent Assoc. 2015 Apr;146(4):233-40. doi: 10.1016/j.adaj.2014.12.014. PMID 25819654
- [Derived] de Geus JL, de Lara MB, Hanzen TA, Fernandez E, Loguercio AD, Kossatz S, Reis A. One-year follow-up of at-home bleaching in smokers before and after dental prophylaxis. J Dent. 2015 Nov;43(11):1346-51. doi: 10.1016/j.jdent.2015.08.009. Epub 2015 Aug 21. PMID 26303401